CLINICAL TRIAL: NCT04675307
Title: Multimodal, Task-Aware Movement Assessment and Control: Clinic to the Home
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Boston University (Other)
Responsible Party: Principal Investigator, David Levine, David Levine, MD, MPH, MA- Principle Investigator, Brigham and Women's Hospital
Other Study IDs: 2020P003474
Record Dates: First submitted 2020-12-08; First posted 2020-12-19 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators seek to construct a novel, multimodal, distributed system that facilitates a new paradigm of home-based medical surveillance and treatment for frail older adults centered on timely diagnosis of movement system impairments and personalized intervention. Measurements from a heterogeneous set of complementary sensors will be combined with clinically-informed and data-learned dynamic models of human motion to enable real-time activity recognition (e.g., sitting, standing, walking) and movement assessments (e.g., speed, repetition, quality). As the study progresses, the system will be integrated with wearable assistive technology to provide "smart", activity-specific assistance of movement deficits or the activation of caregivers if a decline in function is detected. Finally, the investigators will test the combined assessment and intervention system in the clinic and the home, identifying challenges and solutions for the scaling up to unconstrained real-world settings.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Capacity to consent
* Community dwelling
* Ability to follow 3-step commands
* Lives within 15 miles of Boston

Exclusion Criteria:

* Undomiciled
* Active substance use disorder
* Active psychosis
* Domestic violence or neglect
* Inability to communicate with investigators
* Other comorbidities that prevent full participation in the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population will consist of frail adults and frail older adults. Frailty is defined as a state of increased vulnerability and reduced ability to recover after a stressful event, leading to adverse health outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-02-17 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-02 (Estimated)

PRIMARY OUTCOMES:
Video and inertial motion unit capture | 1 recording episode, approximately 3 hours
  Successfully capture video and inertial motion unit capture of subjects as they perform various movement assessments.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States